CLINICAL TRIAL: NCT01359696
Title: An Open-Label, Phase I, Dose Escalation Study Evaluating the Safety, Tolerability, and Pharmacokinetics of GDC-0425 Administered With and Without Gemcitabine in Patients With Refractory Solid Tumors or Lymphoma
Brief Title: A Study Evaluating the Safety, Tolerability, and Pharmacokinetics of GDC-0425 Administered With and Without Gemcitabine in Patients With Refractory Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DPM4957g; GO00767 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2011-05-23; First posted 2011-05-25 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Solid Tumor
Keywords: solid cancers
MeSH Terms: interventions — GDC-0425; Gemcitabine

ARMS (1):
- A (Experimental)
  Interventions: Drug: GDC-0425; Drug: gemcitabine

INTERVENTIONS:
Drug: GDC-0425 — Oral escalating dose
Drug: gemcitabine — Intravenous repeating dose

SUMMARY:
This is an open-label, multicenter, Phase I, dose-escalation study to assess the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of GDC-0425 administered with and without gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1
* Signed Informed Consent Form
* Histologically or cytologically documented, locally advanced or metastatic solid tumors or lymphoma for which standard therapy either does not exist or has proven ineffective or intolerable
* Adequate hematologic and end-organ (liver and kidney) function
* For female patients of childbearing potential and male patients with partners of childbearing potential, agreement by the patient that the patient and/or partner will use an effective form of contraception
* Patients enrolled in certain phases must be willing to provide fresh and/or archival tumor samples

Exclusion Criteria:

* History of prior significant toxicity from a same class of agents as GDC-0425 or gemcitabine requiring discontinuation of treatment
* Allergy, hypersensitivity or contraindication to the GDC-0425 formulation or gemcitabine
* Experimental therapy or anti-cancer therapy within 4 weeks prior to the first dose of study drug treatment
* Radiotherapy within 2 weeks prior to first dose of study drug treatment
* More than two regimens of cytotoxic chemotherapy for the treatment of locally advanced or metastatic cancer
* History of receiving high-dose chemotherapy requiring bone marrow or stem cell support
* History of receiving radiation to more than 25% of bone marrow-bearing areas
* Acute drug-related toxicities from previous therapies have not resolved prior to study entry, except for alopecia and mild neuropathy
* Current severe, uncontrolled systemic disease (including but not limited to clinically significant cardiovascular, pulmonary, or renal disease or ongoing or active infection) excluding cancer
* Significant heart disease and heart dysfunction including but not limited to uncontrolled severe hypertension, heart failure, and reduced cardiac contractility
* Uncontrolled ascites, due to diseases other than cancer
* Inability or unwillingness to swallow pills/capsules
* History of malabsorption or other condition that would interfere with drug absorption
* Any history of active stomach and/or intestine bleeding within the 6 months prior to screening
* Known HIV infection
* Pregnancy, lactation, or breastfeeding
* Known brain metastases that are untreated, symptomatic, or require therapy to control symptoms
* Inability to comply with study and follow up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-07-11 (Actual); Primary Completion 2014-05-29 (Actual); Study Completion 2014-05-29 (Actual)

PRIMARY OUTCOMES:
Incidence of all adverse events graded according to NCI CTCAE, v4.0 | Up to 1 year
Incidence of dose limiting toxicities (DLTs) | Up to 35 days
Pharmacokinetic property of GDC-0425: determination of plasma drug concentration | Up to 12 months or early study discontinuation
Pharmacokinetic property of GDC-0425: exposure | Up to 12 months or early study discontinuation
Pharmacokinetic property of GDC-0425: half-life | Up to 12 months or early study discontinuation
Severity of all adverse events graded according to NCI CTCAE, v4.0 | Up to 1 year

SECONDARY OUTCOMES:
Antitumor activity of GDC-0425 in combination with gemcitabine: determination of tumor response using RECIST v1.1 for patients with measurable disease | Up to 12 months or early study discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Chia Portera, M.D., Ph.D., Study Director — Genentech, Inc.
Locations (3):
- United States (2):
  - Karmanos Cancer Institute.., Detroit, Michigan
  - Sarah Cannon Cancer Center, Nashville, Tennessee
- Institut Gustave Roussy; Ser. de Med. Nucleaire; Cancerologie Endo, Villejuif, France